CLINICAL TRIAL: NCT03051334
Title: Changes in Ascending Aorta Size After Transcatheter Aortic Valve Replacement in Severe Bicuspid Aortic Stenosis: A Pilot Study With Echocardiographic Follow-up
Brief Title: Ascending Aortic Dilation in BiAV After TAVR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Kwan Kim, Director, Division of Cardiology, Clinical Professor, Seoul National University Hospital
Other Study IDs: 1701-104-825
Record Dates: First submitted 2017-02-08; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- BiAV: Bicuspid aortic valve
  Interventions: Other: diagnosed as bicuspid aortic valve
- TAV: Tricuspid aortic valve

INTERVENTIONS:
Other: diagnosed as bicuspid aortic valve
  Groups: BiAV

SUMMARY:
This study sought to evaluate changes in ascending aorta size after transcatheter aortic valve replacement (TAVR) in patients with bicuspid aortic valve (BiAV) compared with patients with tricuspid aortic valve (TAV).

DETAILED DESCRIPTION:
The growth rate of ascending aorta was calculated as annual growth rate using baseline and the last echocardiography. The difference in ascending aorta growth rates between the two groups (BiAV and TAV) were analyzed by independent t-test.

ELIGIBILITY:
Inclusion Criteria:

* Severe AS who underwent TAVR

Exclusion Criteria:

* ascending aorta more than 50mm

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Severe AS who underwent TAVR
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2017-12-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
changes in dimension of ascending aorta | baseline and 1year after TAVR
  the annual growth rate of ascending aorta(mm/year) using echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea